CLINICAL TRIAL: NCT03929458
Title: Association of Uremic Sarcopenia and Mitochondrial Copy Number and Its Clinical Correlates in Taiwanese Hemodialysis Patients
Brief Title: Association of Uremic Sarcopenia and Mitochondrial Copy Number and Its Clinical Correlates
Status: Completed | Type: Observational
Sponsor: Tungs' Taichung Metroharbour Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 107061
Record Dates: First submitted 2019-04-22; First posted 2019-04-26 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Sarcopenia; Mitochondrial DNA
Keywords: oxidative stress; Sarcopenia; copy number of mitochondrial DNA (mtDNA)
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Sarcopenia is the decline of muscle mass and strength with age. Evidence suggests that oxidative stress and molecular inflammation play important roles in age-related muscle atrophy. The two factors may interfere with the balance between protein synthesis and breakdown, cause mitochondrial dysfunction, and induce apoptosis. Sarcopenia, inflammation and oxidative stress is highly prevalent in hemodialysis patients and may contribute to mortality. The copy number of mitochondrial DNA (mtDNA) is affected by oxidative stress in blood circulation. This study aimed to test whether mtDNA copy number correlates with oxidative stress and some uremic toxins in nondiabetic hemodialysis(HD) patients. 200 nondiabetic hemodialysis patients and 50 healthy subjects will be enrolled. This study will be performed to investigate quantitative changes in mtDNA occur in HD patients with and without sarcopenia. Copy number of mtDNA in leukocyte DNA is determined by real-time polymerase chain reaction in HD patients and 50 age- and sex-matched control subjects. In addition, correlation of the alterations of albumin redox status, 8-isoprostane, plasma IL-6 ,LBP and TNF-a and as well as various uremic toxins will be performed.

DETAILED DESCRIPTION:
Research design and methods Subjects In this study, we shall recruit 200 patients on maintenance hemodialysis. In addition, 50 age- and sex-matched subjects act as controls. The HD patients have been on stable dialysis for at least 3 months HD patients are being treated three times weekly with standard bicarbonate dialysis (Na 138 mmol/L, HCO3 35 mmol/L, K 1.5 mmol/L, Ca 1.25 mmol/L, Mg 0.75 mmol/L) and by high-flux HD with synthetic membranes (dialysis filters surface area: 1.7 to 2.1 m2). All HD patients enroll in our study will be tested with DEXA and handgrip strength. Demographic data will be collected and laboratory examination are conducted as listed below.

Biochemical Determinations Blood samples for laboratory testing were drawn from the venous end of a vascular access at the beginning of the hemodialysis session and then stored at -80°C until time of analysis. The high sensitive C-reactive protein (hsCRP) levels were determined by a commercial immunoturbidimetric assay using a Hitachi autoanalyzer (model 7170). The detection limit and interval for CRP was 0.1 mg/L and 0.1-500.0 mg/L, respectively. The baseline serum albumin was measured by the bromocresol green method on a Hitachi autoanalyzer (model 7170). Serum levels of cholesterol, triglyceride, and low- and high-density lipoprotein cholesterol were determined by standard laboratory methods.

Determination of relative leucocyte mtDNA copy number The real-time PCR reaction was performed in triplicate for each reaction. The 10ul PCR reaction contains 1X TaqMan Universal PCR Master Mix buffer, 500nM of each primer, 200nM of TaqMan probe, and 0.2-2ng of total genomic DNA extract, PCR conditions are 2 min at 50℃, 10 min at 95℃, followed by 40 cycles of 15 s of denaturation at 95℃ and 60 s of annealing/extension at 60℃. Real-time quantitative analysis was performed on StepOne Real-Time PCR system(ABI). The primers and probes for real-time PCR are listed in Table 1. The PCR products that involve mitochondria DNA(MtDNA) and nuclear DNA.

Standard Curve:

Standard DNA solutions for the mitochondrial genome and the nuclear 18S rRNA dene (nDNA) were generated from PCR products cloned in a vector of pCR2.1-TOPO. Serial dilutions were made and RT-QPCR reactions were performed to construct the standard curve from Ct values and the number of copies of the standard plasmid DNA.

Determination of mtDNA/nDNA Ratio as a measure of mtDNA Content:

The copy number of the mtDNA and the nDNA is calculated using the threshold cycle number (Ct) and intrapolating from the standard curve. The ratio of the copy number of mtDNA to the copy number of nDNA is measurement of mtDNA content.[30] Measurement of the Albumin Redox State Measurement of the albumin redox state was performed using the high-performance liquid chromatography (HPLC) method reported previously [31]. The HPLC-fluorescence detection (HPLC-FD) system consisted of an AS-8010 autosampler (injection volume, 2 mL per specimen; Tosoh, Tokyo, Japan) and a Model FS-8000 fluorescence detector (excitation wavelength, 280 nm; emission wavelength, 340 nm) with a CCPM double-plunger pump (Tosoh) in conjunction with a SC-8020 system controller (Tosoh). A Shodex-Asahipak ES-502N 7C column [Showa Denko, Tokyo, Japan; 10×0.76 cm (inner diameter), dimethylaminoethyl-form for ion-exchange HPLC, column temperature, 35°C±0.5°C] or in some instances two Asahipak GS-520H columns [Asahi Chemical Industry; Kawasaki, Japan; 25×0.75 cm (inner diameter) maintained at 32°C] were used. Linear gradient elution was carried out with an ethanol level increasing from 0% to 5% in 0.05 M sodium acetate and 0.40 M sodium sulfate buffer (pH 4.85; acetate-sulfate buffer) at a flow rate of 1.0 mL/min. Deaeration of the buffer solution was performed by helium bubbling. Based on the HPLC profiles of HSA obtained from these procedures, the values for each fraction were subjected to numerical curve fitting, and the fractions of HMA, HNA-1, and HNA-2 to total HSA were calculated.

Measurements of Liposaccharide-binding protein (LBP) The LBP was determined from serum samples and controls using standardized enzymelinked immunosorbent assay (ELISA) methods, and serum from normal control subjects was used for interassay variation.

Total of 8-iso-PGF2-alpha Analysis Total 8-iso-PGF2-alpha concentrations in plasma were measured by a specific enzyme immunoassay (EIA) kit (Cayman Chemical, Ann Arbor, Mich). Samples were centrifuged and the supernatants were collected, purified as stated previously and stored at -80°C until assayed. Samples were assayed at 50 μl after a 1:10 or 1:20 dilution and read at 420 nm in a 96 well microplate reader. The assay has been validated to obtain a high correlation (0.95) between added known amounts of 8-isoprostane and the concentration measured by EIA and has been directly validated by gas chromatography/mass spectrometry. The antiserum used in this assay has a 100%cross reactivity with 8-iso-PGF2-alpha 0.2% each with PGF2-alpha, PGF3, PGE1, PGE2, 0.1% each with 6-keto-PGF1-alpha. The detection limit of the assay is 4 pg/ml and the range of standard curve was from 3.9 to 500 pg/ml.

Measurements of Serum total p-cresol and Indoxyl sulfate Plasma concentrations of total p-cresol sulfate(PCS) and indoxyl sulfate( IS) are analyzed with High-performance liquid chromatography (HPLC). Briefly, for binding competition, 200μl serum to which we added 20μl 0.50mM 1-naphthalenesulfonic acid (internal standard) was vortex-mixed with 250μl 0.24M sodium octanoate (binding competitor).After incubation at room temperature for 5min, we added 2ml cold acetone to precipitate proteins. Following vortex-mixing and centrifuging at 4 ◦C, 1860×g for 20 min, the supernatant was transferred to 12mm×100mm, GL 14 glass test tubes and 2ml dichloromethane was added. After vortex-mixing and centrifuging at 4 ◦C, 1860×g for 10min, 200μl of the upper layer was transferred to glass autosampler vials, followed by addition of 20μl 1M HCl and 15μl was injected onto the HPLC. The HPLC analysis was performed on an Agilent 1100 series LC (Santa Clara, CA), and Agilent ChemStations software were used for the chromatographic analysis. The separation was carried out on a ZORBAX SB-C18 Solv Saver Plus HPLC column (5 μm, 3.0 mm×150 mm).at a flow rate of 0.6 ml/min. Mobile phase A is 0.2% trifluoroacetic acid in Milli-Q water and mobile phase B is 0.2% trifluoroacetic acid in acetonitrile. The analytical method consists of an isocratic run with 92% mobile phase A for 23 min.. Each analytical run was followed by a 1.3 min washout gradient to 100% B. Column temperature was 25 ◦C, and autosampler tray temperature was 6 ◦C. We quantified the analytes by using the analyte to standard peak area ratio on a Agilent 1100 High Performance Fluorescence detector G1321A. Detector settings were λex 260 nm/λem288nm for p-cresyl sulfate and λex 280 nm/λem 390nm for indoxyl sulfate and internal standard. Quantitative results are obtained and calculated in terms of their concentrations (mg/L).

Handgrip strength Muscle strength is assessed in the dominant hand using a Jamar hand dynamometer (Lafayette Instrument Company, USA). Patients are ﬁrst familiarized with the device and were then examined standing with both arms extended sideways from the body with the dynamometer facing away from the body. Patients were instructed to grip the dynamometer with the maximum strength in response to a voice command, and the highest value of three measurements was considered for the study. Handgrip strength (HGS) values under the 30th percentile (Table 2) from a speciﬁc-population reference value adjusted for age and sex were considered as reduced [32].

Dual-Energy X-ray Absorptiometry (DEXA) DEXA is a widely used reference method for body FFM and FM measurements.10 DEXA was performed using a Lunar Prodigy (GE Medical Systems, Madison, WI). Whole-body scans were performed according to manufacturer's instructions, and body FM (FMDEXA), LTM (LTMDEXA) and bone mineral content are analyzed using the manufacturer's software. The DEXA method uses an X-ray tube with a filter to generate low-energy (40 kV). and high-energy (70 or 100 kV) photons. When photonsat different energy levels pass through tissue, their absorptions can be expressed as a ratio of attenuation at lower or higher energy levels. DEXA estimate of FFM was calculated as a sum of LTM and bone mineral content estimates.

All patients will be examined by the same observer. Overall, AWGS recommends using 2 standard deviations below the mean muscle mass of young reference group or the lower quintile as the cutoff value determination. Moreover, AWGS recommends using height-adjusted skeletal muscle mass instead of weight-adjusted skeletal muscle mass, and the suggested cutoff values were 7.0 kg/m2 in men and 5.4 kg/m2 in women by using DEXA.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes aged between 20-90 years.
* Received stable hemodialysis at least 3 months.
* Written informed consent.

Exclusion Criteria:

* patients with severe infections, severe heart disease and liver disease, malignancy, autoimmune disorders, severe malnutrition, or clinical conditions requiring oral nutrition supplements;
* Inability to follow protocol.
* Pregnancy or wishing/trying to get pregnant

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients have to be at least 20-years-old and on outpatient hemodialysis (HD) for at least 3 months.
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2019-05-07 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Determination of mtDNA/nDNA Ratio as a measure of mtDNA Content | 1 years
  The copy number of the mtDNA and the nDNA is calculated using the threshold cycle number (Ct) and intrapolating from the standard curve. The ratio of the copy number of mtDNA to the copy number of nDNA is measurement of mtDNA content.

SECONDARY OUTCOMES:
Plasma uremic toxins analysis | 1 years
  ndoxyl sulfate (IS) and para-cresol (p-cresol) belong to the group of protein-bound uremic toxins that are poorly cleared by dialysis and are associated with poor clinical outcomes.the group of protein-bound uremic toxins that are poorly cleared by dialysis and are associated with poor clinical outcomes.
Total of 8-iso-PGF2-alpha Analysis | 1 years
  Total 8-iso-PGF2-alpha concentrations in plasma were measured by a specific enzyme immunoassay (EIA) kit
Analysis of biomarkers of IL-6 | 1 years
  The IL-6 was determined from serum samples and controls using standardized enzymelinked immunosorbent assay (ELISA) methods
Analysis of biomarkers of TNF-α | 1 years
  The TNF-α was determined from serum samples and controls using standardized enzymelinked immunosorbent assay (ELISA) methods
Analysis of biomarkers of Liposaccharide-binding protein (LBP) | 1 years
  The LBP was determined from serum samples and controls using standardized enzymelinked immunosorbent assay (ELISA) methods
Measurement of the Albumin Redox State | 1 years
  the fractions of HMA, HNA-1, and HNA-2 to total HSA were measured using HPLC

CONTACTS AND LOCATIONS:
Overall Officials: Paik Seong Lim, PhD, Principal Investigator — Tungs' Taichung Metroharbour Hospital
Locations (1):
- Tungs' Taichung MetroHarbour Hospital, Taichung, Taiwan